CLINICAL TRIAL: NCT03687632
Title: A Phase 2 Open Label Trial of ST266 Eye Drops in the Treatment of Persistent Corneal Epithelial Defects
Brief Title: ST266 Eye Drops for the Treatment of Persistent Corneal Epithelial Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST266-PED-201
Record Dates: First submitted 2018-09-24; First posted 2018-09-27 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Persistent Corneal Epithelial Defect

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, open label trial to determine if treatment with ST266 eye drops for 28 days heals the study eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm - active (Experimental): ST266 eye drops given to the study eye for 28 days (112 doses total will be administered).
  Interventions: Biological: ST266

INTERVENTIONS:
Biological: ST266 — 1X ST266 applied in a dose of one drop (30-50 µL) in the study eye for 28 days (112 doses total will be administered).

SUMMARY:
The primary aim of the study is to evaluate the clinical response of ST266 treated subjects with persistent corneal epithelial defects during 28 days of therapy. The secondary endpoint is the response rate within 14 days of treatment.

DETAILED DESCRIPTION:
Efficacy:

The primary aim of the study is to evaluate the clinical response of ST266 treated subjects with persistent corneal epithelial defects during 28 days of therapy. The secondary endpoint is the response rate within 14 days of treatment. Failures are subjects that do not completely heal during 28 days of therapy. The epithelial defect can be of any size as long as it is measurable by slit lamp. The longest measurement and the measurement perpendicular to that will be determined and the area calculated. The change in area and perimeter of epithelial defect from baseline through Day 15 (14 days of treatment) and Day 29 (28 days of treatment) will be calculated for each subject. The time to complete re-epithelialization is defined as the time from the start of therapy (Baseline Visit/Day 1) to the Day when no defect is observed. The number and percent of responders and failures will be summarized at each visit. Graphical representation of percent of responders and failures will be provided. The change in area and perimeter of epithelial defect from baseline through Day 15 (14 days of treatment) and Day 29 (28 days of treatment) will be summarized. Visualization of mean (Standard Deviation) of the change in area and perimeter will be provided at each time point. The time to complete re-epithelialization will be summarized and listed.

Safety:

Subject demographics, baseline characteristics and relevant medical history will be summarized and listed. Data for ST266 administration and concomitant therapies will be listed.

The number and percent of subjects with treatment emergent adverse events and ST266 related adverse events will be tabulated by system organ class and preferred terms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 years and over.
* Subjects with a PED present for at least seven (7) days.
* The defect may be of any size and must be measurable by slit lamp.
* In the Investigator's opinion, the defect is persistent i.e., the defect has not shown improvement despite conventional treatment such as tear supplements and bandage contact lenses.
* The original defect to the cornea must be the result of any injury, infection, disease or surgery to the eye.

Exclusion Criteria:

* Subjects currently being treated with cenegermin.
* Subjects who require treatment with autologous serum eyedrops throughout the duration of the trial. If, in the opinion of the investigator, autologous serum eyedrop treatment can be safely stopped, the subject may be included in the clinical trial.
* Subjects who require treatment with other amnion products throughout the duration of the trial. If, in the opinion of the investigator, the amniotic product treatment can be safely stopped, the subject may be included in the clinical trial.
* Subject who requires treatment with amniotic membrane throughout the duration of the trial. If the amniotic membrane can be safely stopped, the subject may be included in the clinical trial. Note: The amniotic membrane must be removed at least one (1) day prior to the baseline visit.
* Subjects who require treatment with bandage contact lens that cannot be removed at least 24 hours prior to screening. If the bandage contact lens can be safely removed, the subject may be included in the clinical trial.
* Subject with an uncontrolled lid or ocular infection.
* History of alkali burns of the cornea.
* The circumference affected by limbal blood vessel ischemia is greater than 75 percent of the circumference.
* Subjects with severe lid abnormalities contributory to the persistence of the PED such as the inability to close the lids.
* Subjects who have a history of AIDS or HIV.
* Treatment with systemic corticosteroids (equivalent to >10 mg/day of prednisone) or immunosuppressive (including Plaquenil) or chemotherapeutic agents within 7 days prior to Day 1, or likely to receive one of these therapies during study participation.
* Subjects who have participated in a clinical trial within 30 days prior to Day 1.
* Subjects who have more than one distinct PED in the study eye prior to screening visits. Subjects who develop PEDs after the screening visit will remain in the study; however, only the original study PED will be assessed.
* Subjects with bullous keratopathy.
* Subjects with corneal perforation or impending corneal perforation.
* For subjects with bilateral PEDs, only the eye with the larger PED should be entered in to the study. The non-study eye will receive standard of care treatment and will be observed throughout the trial.
* Female subjects who are pregnant or breastfeeding. Female subjects who are neither postmenopausal nor surgically sterile require a negative urine pregnancy test on Day 1 visit.
* Epithelial defect was classified as a progressive corneal melt caused by an immunological process such as rheumatoid melt or Mooren's ulceration.
* Subjects with recurrent corneal erosion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with complete healing of PED during 28 days of treatment starting | 28 days
  Healing is defined as the complete re-epithelialization of the epithelial defect as determined by slit lamp examination with fluorescein staining.

SECONDARY OUTCOMES:
Safety endpoint of the incidence of adverse and serious adverse events | 28 days
  The secondary safety endpoint is the incidence of adverse and serious adverse events throughout the 28 days of treatment. For the safety evaluation, changes in visual acuity, IOP, and fluorescein staining will be considered as safety measures.
Percent of subjects with complete healing within 14 days of starting treatment | 14 days
  Healing is defined as the complete re-epithelialization of the epithelial defect as determined by slit lamp examination with fluorescein staining.
Time (in days) to complete re-epithelialization of the study eye | This assessment will occur during clinic visits on days 4, 8, 11, 15, 22 and 29.
  Re-epithelialization of the epithelial defect as determined by slit lamp examination with fluorescein staining.
Persistence of complete corneal re-epithelialization in the study eye | The measurement will be made 7 days after end of treatment (at end of study visit).
  Corneal re-epithelialization in the study eye as determined by whether the healed epithelium remains intact after complete re-epithelialization is confirmed in the study eye, as determined by slit lamp examination with fluorescein staining.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Price Vision Group, Indianapolis, Indiana
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Univesity of Pittsburgh, Pittsburgh, Pennsylvania
  - University of West Virginia, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No